CLINICAL TRIAL: NCT04509518
Title: The Effectiveness of Selected Physical Therapy Exercise Program With or Without Transcutaneous Electrical Nerve Stimulation on Male Patients With Pudendal Neuralgia
Brief Title: Effectiveness of Selected Physical Therapy Exercise Program and Transcutaneous Electrical Nerve Stimulation on Patients With Pudendal Neuralgia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Marwa Eid, assistant professor of physical therapy for surgery, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PN
Record Dates: First submitted 2020-08-09; First posted 2020-08-12 (Actual); Last update posted 2020-08-12 (Actual); Status verified 2020-08

CONDITIONS: Pudendal Neuralgia
MeSH Terms: conditions — Pudendal Neuralgia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (Experimental): Participants in the study group received exercise therapy program plus additional TENS therapy
  Interventions: Other: Exercise therapy program plus TENS therapy
- Control group (Other): Participants in the study group received exercise therapy program plus sham TENS
  Interventions: Other: Exercise therapy program plus TENS therapy

INTERVENTIONS:
Other: Exercise therapy program plus TENS therapy — All patients were receiving the same physical therapy exercise program, 3 times per week for 12 weeks in the form of pelvic floor relaxation exercises, diastasis correction exercises , myofascial trigger points release, connective tissue manipulation and progressive abdominal strengthening exercises. Pelvic floor relaxation exercises included pelvic floor release stretches, Proprioceptive Neuromuscular Facilitation technique, and pelvic floor drop exercises in addition to TENS therapy The standard protocol for TENS therapy in this group was 20 minutes of 100 Hz frequency, pulse duration of 200 µsec, three times a week for successive 12 weeks

SUMMARY:
To study the efficacy of adding Transcutaneous Electrical Nerve Stimulation (TENS) to selected physical therapy exercise program on pain in patients with pudendal neuralgia.

Fifty-two male participants with chronic pudendal neuralgia (30-50 years) shared in this study.

Methods: patients were assigned randomly into two groups equal in number; study and control groups with 26 patients in each. All patients were receiving the same physical therapy exercise program, in addition to the same prescribed analgesic medication. Patients in the study group received additional TENS therapy and those in the control group received sham TENS. Treatment was provided three sessions per week for twelve successive weeks. The participants underwent baseline and post treatment assessment for pain level as measured by three methods; Serum Cortisol Level (SCL), Daily Etodolac intake dose (DEID), and Numerical Pain Rating Scale (NPRS).

ELIGIBILITY:
Inclusion Criteria:

* Nonsmoking male patients
* Diagnosed as having unilateral pudendal nerve entrapment resulting in pudendal neuralgia
* Ages ranged between 30 to 50 years
* Did not have any behavioral or cognitive impairments that could prevent them from following simple verbal commands or instructions during tests and training.

Exclusion Criteria:

* Those who had history of skin malignancy
* Diabetes
* Sensory disorders
* Circulatory insufficiency
* Acute infection of the treatment area
* Renal failure
* Myocardial infarction
* Communication problems, or those with pace maker

Ages: 30 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2018-02-10 (Actual); Primary Completion 2019-04-05 (Actual); Study Completion 2019-12-07 (Actual)

PRIMARY OUTCOMES:
Neumerical rating scale | 12 weeks
  It is composed of a numeric segmented horizontal line ranging from 0 which represents "no pain" and 10 which represents "worst imaginable pain"conditions tend to have higher values

CONTACTS AND LOCATIONS:
Locations (1):
- Marwa Eid, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes